CLINICAL TRIAL: NCT02960893
Title: A Phase IIb/III, Randomized, Double-blind, Placebo-controlled Trial of Troriluzole in Adult Participants With Spinocerebellar Ataxia
Brief Title: Trial in Adult Participants With Spinocerebellar Ataxia (SCA)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV4157-201
Expanded Access: NCT06034886 (Available)
Record Dates: First submitted 2016-11-04; First posted 2016-11-10 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Spinocerebellar Ataxias; Spinocerebellar Ataxia Genotype Type 1; Spinocerebellar Ataxia Genotype Type 2; Spinocerebellar Ataxia Genotype Type 3; Spinocerebellar Ataxia Genotype Type 6; Spinocerebellar Ataxia Genotype Type 7; Spinocerebellar Ataxia Genotype Type 8; Spinocerebellar Ataxia Genotype Type 10
Keywords: Spinocerebellar Ataxia; SCA
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Troriluzole - Randomization Phase (Experimental): Troriluzole - Randomization Phase: Participants received Troriluzole 140 mg capsules orally once daily (QD) for 8 weeks.
  Interventions: Drug: Troriluzole
- Placebo - Randomization Phase (Placebo Comparator): Placebo - Randomization Phase: Participants received matching placebo capsules orally QD for 8 weeks.
  Interventions: Drug: Placebo
- Troriluzole/Troriluzole - OLE (Open Label Extension) Phase (Experimental): Participants received Troriluzole 140 mg capsules orally QD for 48 weeks in the extension period and were allowed to participate in 288 weeks for expanded extension phase, for a total of 336 weeks of open-label treatment.
  Interventions: Drug: Troriluzole
- Placebo/Troriluzole - OLE Phase (Experimental): Participants who received placebo during randomization phase, received Troriluzole 140 mg capsules orally QD for 48 weeks in the extension period and were allowed to participate in 288 weeks for expanded extension phase, for a total of 336 weeks of open-label treatment.
  Interventions: Drug: Placebo; Drug: Troriluzole

INTERVENTIONS:
Drug: Troriluzole — Randomization Phase: Neat (i.e., drug substance without excipients); loose filled capsule.
  Arms: Troriluzole - Randomization Phase; Troriluzole/Troriluzole - OLE (Open Label Extension) Phase
Drug: Placebo — Drug: Placebo Randomization Phase: Matching placebo loose filled capsule.
  Arms: Placebo - Randomization Phase; Placebo/Troriluzole - OLE Phase
Drug: Troriluzole — OLE phase: Neat capsule or formulated capsule (i.e., drug substance with excipients).
  Arms: Placebo/Troriluzole - OLE Phase; Troriluzole/Troriluzole - OLE (Open Label Extension) Phase

SUMMARY:
The primary purpose of this study was to compare the efficacy of BHV-4157 (Troriluzole) 140 milligrams (mg) once daily versus placebo after 8 weeks of treatment in participants with spinocerebellar ataxia (SCA).

DETAILED DESCRIPTION:
The study was conducted in 2 phases: Randomization Phase (8 weeks) followed by an open-label Extension Phase (336 weeks). During the Randomization Phase, participants received either Troriluzole 140 mg or matching placebo up to 8 weeks. Participants who agreed to enter the Open-label Extension Phase continued dosing of Troriluzole 140 mg for 336 weeks. The study was subsequently amended to follow participants for a total of 336 weeks in the Open-label Extension Phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with a known or suspected diagnosis of the following specific hereditary ataxias: SCA1, SCA2, SCA3, SCA6, SCA7, SCA8 and SCA10
* Ability to ambulate 8 meters without assistance (canes and other devices allowed)
* Screening total Scale for the Assessment and Rating of Ataxia (SARA) score ≥8
* Score of ≥ 2 on the gait subsection of the SARA
* Determined by the investigator to be medically stable at baseline/randomization and must be physically able and expected to complete the trial as designed

Key Exclusion Criteria:

* Any medical condition other than one of the hereditary ataxias specified in the inclusion criteria that could predominantly explain or contribute significantly to the participants symptoms of ataxia
* Mini Mental State Exam (MMSE) score < 24
* SARA total score of > 30 points at screening
* Clinical history of stroke
* Active liver disease or a history of hepatic intolerance to medications that in the investigator's judgment, is medically significant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - CNS Trial, Long Beach, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University (Massachusetts General Hospital), Boston, Massachusetts
  - Harvard University (Beth Israel Deaconess Medical Center), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Texas Southwestern, Dallas, Texas
  - Houston Methodist Research Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmahmann JD, Pierce S, MacMore J, L'Italien GJ. Development and Validation of a Patient-Reported Outcome Measure of Ataxia. Mov Disord. 2021 Oct;36(10):2367-2377. doi: 10.1002/mds.28670. Epub 2021 Jun 11. PMID 34115419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 181 participants were screened, and 141 of these participants were randomized to treatment at 18 sites in the United States.
Groups:
- Troriluzole - Randomization Phase: Participants received Troriluzole 140 milligrams (mg) capsules orally once daily (QD) for 8 weeks.
- Placebo - Randomization Phase: Participants received matching placebo capsules orally QD for 8 weeks.
- Troriluzole/Troriluzole - Open Label Extension (OLE) Phase: Participants received Troriluzole 140 mg capsules orally QD for 48 weeks in the extension period and were allowed to participate in 288 weeks for expanded extension phase, for a total of 336 weeks of open-label treatment.
Period: Randomization Phase (8 Weeks)
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Troriluzole/Troriluzole - Open Label Extension (OLE) Phase | Placebo/Troriluzole - OLE Phase
Started | 71 | 70 | 0 | 0
Completed (Completed the Randomization Phase) | 64 | 68 | 0 | 0
Not Completed | 7 | 2 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0
Not completed — Withdrawal by Participant | 2 | 1 | 0 | 0
Not completed — Reason Not Specified | 0 | 1 | 0 | 0
Period: Open Label Extension Phase (336 Weeks)
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Troriluzole/Troriluzole - Open Label Extension (OLE) Phase | Placebo/Troriluzole - OLE Phase
Started | 0 | 0 | 64 | 67 (One participant in placebo arm who completed Randomization Phase did not continue to OLE Phase)
Completed | 0 | 0 | 28 | 36
Not Completed | 0 | 0 | 36 | 31
Not completed — Adverse Event | 0 | 0 | 4 | 4
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 3
Not completed — Physician Decision | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 19 | 18
Not completed — Sponsor Request | 0 | 0 | 4 | 2
Not completed — Miscellaneous | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (Randomization Phase): All participants who received at least one dose of study drug during the Randomization Phase.
Groups:
- Troriluzole - Randomization Phase: Participants received Troriluzole 140 mg capsules orally once daily (QD) for 8 weeks.
- Placebo - Randomization Phase: Placebo - Participants received matching placebo capsules orally QD for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (15.08) | 51.6 (13.74) | 52.1 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 36 | 33 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 65 | 64 | 129
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 11 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 56 | 53 | 109
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 2 | 5
Spinocerebellar Ataxia (SCA) Genotype [Count of Participants; unit: Participants] — The Spinocerebellar Ataxia (SCA) data displayed are not grades or stages of disease, but rather the SCA genotypes, which do not correlate with severity of disease.
  Participants
    SCA1 | 17 | 18 | 35
    SCA2 | 19 | 18 | 37
    SCA3 | 8 | 6 | 14
    SCA6 | 16 | 15 | 31
    SCA7 | 2 | 5 | 7
    SCA8 | 6 | 6 | 12
    SCA10 | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score on the Scale for the Assessment and Rating of Ataxia (SARA) at Randomization Phase Week 8
Description: The severity of ataxia was assessed with the SARA, an 8-item clinical rating scale from 0 (no ataxia) to 40 (most severe ataxia). The total score was derived as the sum of the individual items, which included gait (0-8), stance (0-6), sitting (0-4), speech disturbance (0-6), finger chase (0-4), nose-finger test (0-4), fast alternating hand movements (0-4), and heel-shin slide (0-4). Since the finger chase, nose-finger test, fast alternating hand movements, and heel-shin slide were repeated on both the right and left side, the average of the right and left side assessments was used to derive the total score. A negative change in score shows improvement.
Time Frame: Baseline, Randomization Phase Week 8
Population: Full Analysis Set (FAS): All randomized participants with at least one dose of study drug and a baseline and post-baseline Total SARA score during the Randomization Phase. Here, number of participants analyzed signifies the number of evaluable participants with change from baseline in Total SARA score at Week 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Troriluzole - Randomization Phase: Participants received Troriluzole 140 mg capsules orally QD for 8 weeks.
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 63 | 68
score on a scale | -0.810 (1.7653) | -1.059 (2.3221)
Statistical Analysis 1: Comparison: Troriluzole - Randomization Phase vs Placebo - Randomization Phase; Test type: Superiority; p = 0.519, Mixed Model with Repeated Measures — Significance was evaluated at a 2-sided alpha level of 0.05; Fixed effects: treatment, baseline (BL) gait severity, visit, treatment-by-visit interaction; Covariate: BL Total SARA score; Random effect: subject; LS Mean = 0.2, 95% CI 2-sided [-0.5 to 0.9], Standard Error of Mean 0.4

2. Secondary Outcome: Number of Participants With Deaths, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Treatment-Emergent AEs (TEAEs) During the Randomization Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition, unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. An SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or suspected transmission of an infectious agent, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes. TEAEs were defined as those AEs that developed, worsened, or became serious after the first dose of study drug.
Time Frame: From first dose of study drug to 30 days post the last dose in the Randomization Phase (Up to 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 71 | 70
Participants
  Deaths | 0 | 0
  SAEs | 4 | 1
  Discontinued due to AEs | 3 | 0
  TEAEs | 40 | 35

3. Secondary Outcome: Number of Participants With Deaths, SAEs, AEs Leading to Discontinuation and TEAEs During the OLE Phase
Description: as for outcome 2
Time Frame: From first dose of study drug to 30 days post the last dose in the OLE Phase (Up to 340 weeks)
Population: Safety Analysis Set (OLE Phase): All participants who received at least one dose of study drug during the OLE Phase.
Measure: Count of Participants; unit: Participants
Groups:
- Troriluzole/Troriluzole - OLE Phase; Placebo/Troriluzole - OLE Phase: Participants received Troriluzole 140 mg capsules orally QD for 336 weeks.
Arm/Group | Troriluzole/Troriluzole - OLE Phase | Placebo/Troriluzole - OLE Phase
Number analyzed (Participants) | 64 | 67
Participants
  Deaths | 2 | 1
  SAEs | 11 | 9
  Discontinued due to AEs | 9 | 4
  TEAEs | 60 | 59

4. Secondary Outcome: Number of Participants Who Received At Least One Dose of Troriluzole in the Randomization Phase or OLE Phase With Deaths, SAEs, AEs Leading to Discontinuation and TEAEs
Description: as for outcome 2
Time Frame: From first dose of study drug to 30 days post the last dose in the OLE Phase (Up to 348 weeks after last randomization participant was enrolled)
Population: All participants who received at least one dose of Troriluzole during the Randomization Phase or OLE Phase.
Measure: Count of Participants; unit: Participants
Groups:
- Troriluzole - Overall: Participants received at least one dose of Troriluzole 140 mg capsule orally QD during the Randomization Phase or OLE Phase.
Arm/Group | Troriluzole - Overall
Number analyzed (Participants) | 138
Participants
  Deaths | 3
  SAEs | 23
  Discontinued due to AEs | 19
  TEAEs | 126

5. Secondary Outcome: Number of Participants With Impression of Benefit Via Use of the Patient Global Impression of Change (PGI-C) Index Scale During Randomization Phase
Description: PGI-C is a patient self-reported global index scale that was used to rate the response of a condition to therapy. Participants rated their impression of benefit based on the following 7 categories: No change (or condition has gotten worse); Almost the same, hardly any change at all; A little better, but no noticeable change; Somewhat better, but the change has not made any real difference; Moderately better, and a slight but noticeable change; Better and a definitive improvement that has made a real and worthwhile difference; A great deal better and a considerable improvement that has made all the difference.
Time Frame: Randomization Phase Week 8
Population: Full Analysis Set (FAS): All randomized participants with at least one dose of study drug and a baseline and post-baseline Total SARA score during the Randomization Phase. Here, number of participants analyzed signifies the number of evaluable participants for PGI-C index at Week 8.
Measure: Count of Participants; unit: Participants
Groups:
- Troriluzole - Randomization Phase: Participants received Troriluzole 140 mg capsules orally once daily QD for 8 weeks.
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 63 | 66
Participants
  No Change | 31 | 27
  Almost the same | 15 | 15
  A little better | 7 | 11
  Somewhat better | 3 | 2
  Moderately better | 3 | 7
  Better | 4 | 4
  A great deal better | 0 | 0

6. Other Pre Specified Outcome: Change From Randomization Baseline in Total Score on the SARA at Extension Phase Week 48
Description: as for outcome 1
Time Frame: Randomization Baseline, Extension Phase Week 48
Population: Full Analysis Set (FAS): All randomized participants with at least one dose of study drug and a baseline and post-baseline Total SARA score during the Randomization Phase. Here, number of participants analyzed signifies the number of evaluable participants with change from Randomization baseline in Total SARA score at Week 48.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Troriluzole - Extension Phase: Participants received Troriluzole 140 mg capsules orally QD for 48 weeks.
Arm/Group | Troriluzole - Extension Phase
Number analyzed (Participants) | 96
score on a scale | -0.42 (2.522)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days post the last dose in the OLE Phase (Up to 348 weeks after last randomization participant was enrolled)
Description: Safety Analysis Set: All participants who received at least one dose of study drug during the Randomization Phase/OLE Phase
  MedDRA versions used: Randomization phase: v19.0, OLE Phase: v20.0 and v27.0
Groups:
- Troriluzole/Troriluzole - OLE Phase: Participants received Troriluzole 140 mg capsules orally QD for 48 weeks in the extension period and were allowed to participate in 288 weeks for expanded extension phase, for a total of 336 weeks of open-label treatment.
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Troriluzole/Troriluzole - OLE Phase | Placebo/Troriluzole - OLE Phase
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/70 | 2/64 | 1/67
Serious Adverse Events (participants affected / at risk) | 4/71 | 1/70 | 11/64 | 9/67
Other Adverse Events (participants affected / at risk) | 22/71 | 18/70 | 48/64 | 50/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=71) | Placebo - Randomization Phase (N=70) | Troriluzole/Troriluzole - OLE Phase (N=64) | Placebo/Troriluzole - OLE Phase (N=67)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ankle operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=71) | Placebo - Randomization Phase (N=70) | Troriluzole/Troriluzole - OLE Phase (N=64) | Placebo/Troriluzole - OLE Phase (N=67)
Nausea (Gastrointestinal disorders) | 4 | 4 | 9 | 7
Fatigue (General disorders) | 6 | 3 | 8 | 10
Fall (Injury, poisoning and procedural complications) | 6 | 2 | 21 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 9 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 7 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 8 | 10
Dizziness (Nervous system disorders) | 8 | 1 | 14 | 6
Headache (Nervous system disorders) | 4 | 4 | 12 | 9
Balance disorder (Nervous system disorders) | 1 | 0 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 7 | 7
Urinary tract infection (Infections and infestations) | 0 | 3 | 4 | 9
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 10 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 3
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 9 | 8
COVID-19 (Infections and infestations) | 0 | 0 | 9 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 7 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 5 | 4
Depression (Psychiatric disorders) | 0 | 0 | 4 | 4
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4
Hypertension (Vascular disorders) | 0 | 0 | 4 | 5
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02960893/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT02960893/SAP_001.pdf